CLINICAL TRIAL: NCT05278494
Title: A Randomized, Placebo-Controlled Study to Evaluate the Efficacy of Perioperative Dextromethorphan Compared to Placebo for the Treatment of Postoperative Pain
Brief Title: Dextromethorphan for Treatment of Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nathanael Heckmann (Other)
Responsible Party: Sponsor-Investigator, Nathanael Heckmann, Assistant Professor, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-22-00191
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextromethorphan (Experimental)
  Interventions: Drug: Dextromethorphan Hydrobromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan Hydrobromide — PO
  Arms: Dextromethorphan
Drug: Placebo — PO
  Arms: Placebo

SUMMARY:
A Randomized, Placebo-Controlled Study to Evaluate the Efficacy of Perioperative Dextromethorphan compared to Placebo for the Treatment of Postoperative Pain

DETAILED DESCRIPTION:
There is extensive preclinical evidence that dextromethorphan has an analgesic effect in patients with pain of traumatic origin. The primary objective is to of this study is to evaluate the efficacy of perioperative dextromethorphan compared to placebo for postoperative pain in patients undergoing total knee arthroplasty (TKA).

This is a single-institution, multi-dose, randomized, placebo-controlled, trial to evaluate the efficacy of perioperative dextromethorphan compared to placebo for postoperative pain in patients undergoing TKA. Male and/or female patients will be randomized to either dextromethorphan treatment group (n = 80) or placebo group (n= 80).

Patients will receive 60 mg oral dextromethorphan (or matching placebo) preoperatively, as well as 30 mg 8- and 16-hours postoperatively.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients Age ≥18 planning to undergo total knee arthroplasty
* ASA classes I - III

Main Exclusion Criteria:

* BMI ≥ 35
* History opioid abuse
* History of intractable vomiting after previous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-op opioid use | 24 hours

SECONDARY OUTCOMES:
Subjective pain | preoperatively and 6, 12, 24, and 48 hours postoperatively
  numeric rating scale (NRS) or visual analog scale (VAS)
Postoperative opioid consumption | at 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Keck School of Medicine of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones IA, Piple AS, Yan PY, Longjohn DB, Gilbert PK, Lieberman JR, Gucev GV, Oakes DA, Ratto CE, Christ AB, Heckmann ND. A double-blinded, placebo-controlled, randomized study to evaluate the efficacy of perioperative dextromethorphan compared to placebo for the treatment of postoperative pain: a study protocol. Trials. 2023 Mar 29;24(1):238. doi: 10.1186/s13063-023-07240-0. PMID 36991450